CLINICAL TRIAL: NCT02886026
Title: Is Outpatient PDD Guided Laser Mediated Destruction of Bladder Tumors (LMD-BT) as Good as Conventional Inpatient PDD Guided Transurethral Tumor Resection in Patients With Low Grade Non-invasive (Ta) Bladder Tumors?
Brief Title: Outpatient PDD Guided Laser Mediated Destruction of Bladder Tumors
Acronym: LaserIII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Gregers Gautier Hermann, Consultant Urologist, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URU06
Record Dates: First submitted 2016-06-21; First posted 2016-09-01 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Bladder Cancer
Keywords: Laser; Bladder cancer; Treatment; Outpatient; TUR-BT
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inpatient TUR-BT (Active Comparator): Transurethral bladder tumor resection in operating theatre as inpatient.
  Interventions: Device: Bladder tumor resection using diathermia
- laser bladder tumor destruction (Experimental): Outpatient laser mediated destruction of bladder tumors (LMD-BT)
  Interventions: Device: Diode laser (980 nm) tumor destruction

INTERVENTIONS:
Device: Bladder tumor resection using diathermia — Conventional bladder tumor resection using diathermia
  Arms: Inpatient TUR-BT
Device: Diode laser (980 nm) tumor destruction — Laser mediated destruction of bladder tumors (LMD-BT)
  Arms: laser bladder tumor destruction

SUMMARY:
This study compare the efficacy of conventional photodynamic (PDD) guided transurethral bladder tumor resection in the operating theatre with outpatient PDD guided laser destruction of bladder tumors through flexible cystoscopes.

DETAILED DESCRIPTION:
A prospective randomized two-part clinical trial comprising patients with recurrent pTa low grade bladder tumors.

Study objectives and purpose:

* 1st Objective: To evaluate whether small pTa bladder tumours can be removed with diode laser in an outpatient department with similar efficacy as by TUR-BT resection in the operating theatre.
* 2nd Objective: To evaluate the patients experience of symptoms during laser treatment in the outpatient department (OPD) using quality of life (QOL) questionnaires (symptom evaluation) and Visual Analog Scale Score (pain evaluation).
* 3rd Objective: To evaluate whether patients prefer standard transurethral bladder tumor resection (TUR-BT) in the operating theatre (OT) or laser treatment in the OPD.
* 4th Objective: To evaluate the safety after laser treatment in the OPD.

Efficacy:

* 1st Endpoint: Proportion of patients with no tumor tissue in the bladder after 4 months and 12 months.
* 2nd Endpoint: Visual Analog Scale Score (pain evaluation) in patients having tumor removed by laser in the OPD.

General urinary problems and QOL one week after the laser treatment. The Danish validated questionnaire (QLQ- BLS24) from EORTC will be used.

* 3rd Endpoint: Patients preference for either OPD laser treatment procedure or TUR-BT in the OT as inpatient procedure.
* 4th Endpoint: Character and severity of adverse events in relation to the outpatient treatment.

Study

Inclusion criteria:

1. Ta low grade bladder tumor recurrences
2. Up to a tumor size of 1,5 cm
3. Up to 6 tumors
4. Eligible patients for TUR-BT

Exclusion criteria:

1. Patients with porphyria
2. Known hypersensitivity to Hexvix® or porfhyrins
3. Use of concomitant anticoagulants as Marevan, Marcoumar, and Pradaxa
4. Dementia
5. Macroscopic hematuria
6. Pregnant or breast feeding women
7. Expected poor compliance estimated by the investigators
8. Patients < 18 years
9. Patients who do not read or understand Danish

ELIGIBILITY:
Inclusion Criteria:

1. Ta low grade bladder tumor recurrences
2. Up to a tumor size of 1,5 cm
3. Up to 6 tumors
4. Eligible patients for TUR-BT in GA

Exclusion Criteria:

1. Patients with porphyria
2. Known hypersensitivity to Hexvix® or porfhyrins
3. Use of concomitant anticoagulants as Marevan, Marcoumar, and Pradaxa
4. Dementia
5. Macroscopic hematuria
6. Pregnant or breast feeding women
7. Expected poor compliance estimated by the investigators
8. Patients < 18 years
9. Patients who do not read or understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence histological identified in biopsy obtained during cystoscopy | 4 months
  Numbers (%) of patients vith histological proven recurrence of bladder tumor after 4 months

SECONDARY OUTCOMES:
Lower urinary symptoms caused by laser treatment. | 2 weeks
  Using the EORTC questionnaire QLQ-BLS24 the extent of symptoms are given on a unique score from 0-100, with 0 being no symptoms and 100 are worst symptoms. Mean and range score in the two arms will be compared statistically.
Side effects to laser treatment. | 2 weeks
  Symptoms measured by one unique score according to the Clavien-Dindo grading system. Mean and range score in the two arms will be compared statistically.
Pain during laser treatment | Evaluated immediately after laser treatment
  The patients record pain on a visual analogue scale of 0-10. Zero corresponds to no pain. Ten correspond to the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gregers G Hermann, DM Sc, Principal Investigator — Department of Urology, Frederiksberg hospital
Locations (1):
- Urological department, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No